CLINICAL TRIAL: NCT03312101
Title: Clinical Trail of Therapeutic Physical Exercise for Lower Limb Overpronation in Rugby Young Players
Brief Title: Exercise Program for Lower Limb Pronation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Gabriel Domínguez-Maldonado, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pornation lower limb
Record Dates: First submitted 2017-09-19; First posted 2017-10-17 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Lower Limb Pronation
Keywords: exercise program
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel asigmanet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): exercise program
  Interventions: Other: exercise program
- Control (No Intervention): observation

INTERVENTIONS:
Other: exercise program — functional exercises consisting of a therapeutic exercise program based on concentric strengthening the gluteal muscles (maximus, medius and minimus) , the tensor fasciae latae muscle and the pyramidal muscle; ischiotibial muscle stretching ; and empowerment in eccentric and stretching of the gastrocnemius muscle, soleus muscle, tibialis posterior muscle and flexor of the big toe muscle,
  Arms: Experimental

SUMMARY:
Introduction: The prevalence of biomechanical alterations in the the lower limbs in school-age children is increasing. The aim of this study is to assess the effectiveness of a therapeutic exercise program in child athletes with lower limb overpronation during gait.

Methods: Relevant databases (PubMed and SCOPUS) were searched. A total of 123 young athletes (aged 9-12 years) will be evaluated. Subjects will be tested biomechanical analysis including all relevant angles, as follows: the Helbing angle, the femorotibial angle, and the Fick angle in both limbs. Subjects will be divided into two groups at random. Children in experimental group will participate in an exercise program for three months. Children in control group will not received treatment for three months. After the study, these children will receive the same treatment as children in experimental group.

DETAILED DESCRIPTION:
Firstly, a biomechanical analysis of gait will be performed at CAMD, using a modular electronic baropodometer (Diagnostic Support Walk®), Milletrix Applicazione MFC® (Diasu, Italia) and a video camera (Diagnostic Support S.R.L., Diasu, Italy). We will measure the parameters characterizing lower limb overpronation. The parameters measured during walking will be: Fick angle, femorotibial angle and Helbing angle. Skin Surface markers on anatomical references were placed to measure femorotibial and Helbing angle. To measure the Fick angle we will take a footprint.

Children in the experimental group will be treated with functional exercises consisting of a therapeutic exercise program based on concentric strengthening the gluteal muscles (maximus, medius and minimus) , the tensor fasciae latae muscle and the pyramidal muscle; ischiotibial muscle stretching ; and empowerment in eccentric and stretching of the gastrocnemius muscle, soleus muscle, tibialis posterior muscle and flexor of the big toe muscle.

The selection of the prescribed exercises will be performed according to the principal activity of different muscles and functional impact on the gait. Previous experiences in implementing this exercises program has shown us positive results after three months of application. That is why this temporary intervention for the period was determined.

Parents of children will be instructed to monitor the exercises. They will be given a timetable for controlling autonomous treatment sessions, as well as the dates of the revisions with the evaluator. These reviews will be conducted every 15 days, analyzing the evolution of musculoskeletal disorders, and, if necessary, modifications will be applied in the exercise program.

After three months, a new evaluation will be performed in the same manner as the initial assessment. The purpose of this evaluation is to determine the existence or not of changes in biomechanical parameters studied due the exercices program application.

ELIGIBILITY:
Inclusion Criteria:

* being 9-12 years of age
* having being federated for at least two years (to be a member of the Andalusian Rugby Federation)
* training at least two hours three days a week;
* having lower limb overpronation (Fick angle <12º, femorotibial angle <170º and Helbing angle <175º)

Exclusion Criteria:

* lower limb asymmetry
* biomechanical alteration secondary to an acute disorder

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
lower limb pronation reduction | 3 months
  anthropometric parameters (Fick angle)

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriel Domínguez-Maldonado, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided